CLINICAL TRIAL: NCT00005494
Title: Prospective Study of Health in Runners and Walkers
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 5011; R01HL058621 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-02-29 (Estimated); Status verified 2005-07

CONDITIONS: Coronary Disease; Cardiovascular Diseases; Heart Diseases; Coronary Heart Disease Risk Reduction; Breast Neoplasms; Neoplasms
MeSH Terms: conditions — Coronary Disease; Cardiovascular Diseases; Heart Diseases; Breast Neoplasms; Neoplasms

SUMMARY:
To compare rates of coronary heart disease (CHD), cancer, total mortality and exercise injuries in 68,000 runners and 68,000 walkers during four years of surveillance

DETAILED DESCRIPTION:
BACKGROUND:

Current government physical fitness guidelines state that: 1) the majority of the health benefits from physical activity can be obtained by walking two miles briskly on most days of the week; and 2) the health benefits of physical activity depend principally on the total amount of activity rather than the intensity of the activity. Nevertheless, there are currently no prospective epidemiological studies extant, designed specifically to directly contrast the health benefits and costs of moderate exercise (e.g., walking) versus vigorous exercise (e.g., running).

DESIGN NARRATIVE:

Before the start of the study, 233,000 person-years of follow-up had been accumulated in 56,000 runners (between 1991 and 1997). The runners were resurveyed in 1997 along with 68,000 walkers. The walkers were also solicited through the publication of the questionnaire in Walking magazine followed by a direct mailing of the questionnaire to 425,000 subscribers. Total and cause-specific mortality will be determined from the National Death Index; fatal and nonfatal cancers will be identified from the National Cancer Institute's Surveillance, Epidemiology, and End Results (SEER) and 46 state registries; nonfatal coronary heart disease and injuries will be determined from questionnaires. Survival analyses will be used to test whether runners have greater reduction in heart disease, total mortality, and cancer per unit of exercise. Exercise-related injuries from walking and running will also be examined. Power calculations suggest that detection of differences between runners and walkers, as small as 11% for total mortality, 16% for CHD, 12% for total cancers, and 36% for breast cancer, will be possible. The differences will be adjusted for weekly kilocalories expended by walking and running, for walking and running distance, and for time spent on each activity to test whether these variables account for differences in disease rates between walkers and runners.

By the end of the study, 517,000 person years in 68,000 runners (between 1991 and 2001) will be available for analysis. Survival analysis will be used to test for a dose-response relationship between running mileage and CHD and cancer risk, and whether this relationship is affected by running intensity, running frequency, running history, gender, adiposity, age or medication use. Using conservative rates (25% below published values), statistical power calculations suggest that detectable reduction in coronary heart disease risk as small as 0.71% per mile will be possible, which is far below the estimated reduction from other published studies (2.1%). Additionally, a detectable reduction in breast cancer risk as small as 1.5% per mile run in women is calculated, which is below the 1.7% reduction in risk estimated from other published data.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1998-06; Study Completion 2004-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Williams — University of California Lawrence Berkeley Lab

REFERENCES:
- [Background] Williams PT. Physical fitness and activity as separate heart disease risk factors: a meta-analysis. Med Sci Sports Exerc. 2001 May;33(5):754-61. doi: 10.1097/00005768-200105000-00012. PMID 11323544
- [Background] Williams PT. Health effects resulting from exercise versus those from body fat loss. Med Sci Sports Exerc. 2001 Jun;33(6 Suppl):S611-21; discussion S640-1. doi: 10.1097/00005768-200106001-00030. PMID 11427786
- [Background] Williams PT, Superko HR, Haskell WL, Alderman EL, Blanche PJ, Holl LG, Krauss RM. Smallest LDL particles are most strongly related to coronary disease progression in men. Arterioscler Thromb Vasc Biol. 2003 Feb 1;23(2):314-21. doi: 10.1161/01.atv.0000053385.64132.2d. PMID 12588777
- [Background] Williams PT. The illusion of improved physical fitness and reduced mortality. Med Sci Sports Exerc. 2003 May;35(5):736-40. doi: 10.1249/01.MSS.0000064995.89335.40. PMID 12750581
- [Background] Williams PT, Blanche PJ, Krauss RM. Behavioral versus genetic correlates of lipoproteins and adiposity in identical twins discordant for exercise. Circulation. 2005 Jul 19;112(3):350-6. doi: 10.1161/CIRCULATIONAHA.105.534578. Epub 2005 Jul 11. PMID 16009789